CLINICAL TRIAL: NCT03384797
Title: Blood Biomarker in Early Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00088250
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease
Keywords: blood; biomarker; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers
- Parkinson's Disease

SUMMARY:
Currently, there are no cures or disease modifying therapies for Parkinson's disease (PD). This is partially due to the inability to detect the disease before it has progressed to a stage where there are clinical manifestations. The identification and validation of high throughput biomarkers to measure disease progression (as well as identify pre-clinical disease onset) is critical to the development of disease-modifying or even preventative therapies. In this study, we are testing a blood biomarker for PD. Several detection parameters will be assessed through enrollment of Parkinson's patients and age matched healthy volunteers over 50 years of age to learn more about the analytical process and biological variability.

ELIGIBILITY:
Inclusion

Age matched to PD patient Parkinson's Disease Patients:

* 50 years and older
* PD patient who is seen at the Duke Movement Disorders Center
* Early PD diagnosis (Hoehn and Yahr scale ≤ 3)
* Non-smoking
* No cancer treatment in the last 5 years
* Able to read and speak English

Healthy Control Participants:

* 50 years and older
* Non-smoking
* No cancer treatment in the last 5 years
* Able to read and speak English

Exclusion Criteria:

Parkinson's Disease Patients:

* Known additional neurological disease
* Clinical trial intervention within the last 6 months

Healthy Control Participants:

* Neurological degenerative diseases (such as Parkinson's, Alzheimer's or Huntington's)
* Clinical trial intervention within the last 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients will be recruited from the Duke Movement Disorders Clinic. Healthy adult volunteers will be recruited from the healthy volunteer registry at DEPRU or caregivers of patients seen at the Duke Movement Disorders Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Biological marker of Parkinson's disease | Day 1
  Test for biological marker of Parkinson's disease, mtDNA damage

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Sanders, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Facility, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No